CLINICAL TRIAL: NCT03029936
Title: Obesity-asthma Endophenotype: Assessment of Diaphragm Mobility and Muscle Inflammation Markers in the Adolescence
Brief Title: Obesity-asthma Endophenotype and Diaphragm Mobility in Adolescence
Status: Completed | Type: Observational
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Lui-s Henrique Sarmento Tenorio, Principal Investgator, Universidade Federal de Pernambuco
Other Study IDs: 43599215.4.0000.5208
Record Dates: First submitted 2017-01-19; First posted 2017-01-24 (Estimated); Last update posted 2018-03-19 (Actual); Status verified 2018-03

CONDITIONS: Obesity; Asthma
Keywords: obesity; asthma; diaphragm excursion; pulmonary function test
MeSH Terms: conditions — Obesity; Asthma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Obesity Group
- Asthma Group
- Obesity-Asthma Group
- Control

SUMMARY:
Obesity and asthma share changes that may begin in the fetal development phase. The endophenotype obesity-asthma presents as main characteristic a pattern of inflammatory response different from the habitual Th2 profile of cytokines. In these obese patients, possible changes in the diaphragm muscle can directly influence the dynamics of pulmonary ventilation significantly.

Due to the importance of the diaphragm in pulmonary ventilation, this study will be performed to verify possible alteration in the excursion and diaphragmatic thickness of adolescents with endophenotype obesity-asthma. In parallel, the possible underlying etiopathogenic substrate of this endophenotype will be explored through the dosing of muscle enzymes and inflammatory cytokines and obesity hormones.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents of both sexes, aged 12-21 years;
* For the obesity groups, BMI for gender and age equal to or greater than the 97th percentile;
* Clinical diagnosis of persistent, moderate and severe asthma by a specialist physician and its severity classified according to the GINA (Global Initiative Against Asthma) criteria.

Exclusion Criteria:

* Adolescents with a diagnosis of cardiovascular, rheumatic, osteoarticular, neuromuscular or any other disease that limits the safe performance of the tests proposed by the protocol will be excluded; And those who do not agree to participate in the study.

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 108 adolescents aged 12 years to 21 years will be recruited, of all sexes
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2017-07-30 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Diaphragm mobility | 1 day
  Change in "mm" of diaphragm mobility.

SECONDARY OUTCOMES:
Diaphragm thickness | 1 day
  Change in "cm" of diaphragm thickness.
Th1 Cytokine Levels | 1 day
  Change in "pg/mL" of Th1 Cytokines
Th2 Cytokine Levels | 1 day
  Change in "pg/mL" of Th2 Cytokines

CONTACTS AND LOCATIONS:
Overall Officials: Luis H Tenório, MsC, Principal Investigator — Universidade Federal de Pernambuco
Locations (1):
- Universidade Federal de Pernambuco, Recife, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: No